CLINICAL TRIAL: NCT03473665
Title: Non-Steroidal Anti-inflammatory Drugs in Axial Spondyloarthritis: a Pilot Study
Brief Title: Non-Steroidal Anti-inflammatory Drugs in Axial Spondyloarthritis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Runsheng Wang, MD, MHS, Instructor in Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAR3505
Record Dates: First submitted 2018-03-13; First posted 2018-03-22 (Actual); Results first posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Ankylosing Spondylitis; Axial Spondyloarthritis
Keywords: ankylosing spondylitis; spondyloarthritis
MeSH Terms: conditions — Spondylitis, Ankylosing; Axial Spondyloarthritis; Spondylarthritis | interventions — Indomethacin; Diclofenac; Dacarbazine; Meloxicam; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Indomethacin (Active Comparator): Indomethacin Extended Release Oral Tablet 75mg by mouth, every 12 hours for 6 weeks
  Interventions: Drug: Indomethacin
- Diclofenac (Active Comparator): Diclofenac Delayed Release Oral Tablet 75mg by mouth, every 12 hours for 6 weeks
  Interventions: Drug: Diclofenac
- Meloxicam (Active Comparator): Meloxicam tablet 7.5mg by mouth, every 12 hours for 6 weeks
  Interventions: Drug: Meloxicam
- Celecoxib (Active Comparator): Celecoxib 200mg capsule by mouth, every 12 hours for 6 weeks
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Indomethacin — Indomethacin Extended Release Oral Tablet 75mg every 12 hours for 6 weeks; omeprazole 20mg daily for 6 weeks
  Other Names: INDO; Indomethacin ER
  Arms: Indomethacin
Drug: Diclofenac — Diclofenac Delayed Release Oral Tablet 25mg tablets x 3 tablets every 12 hours for 6 weeks; omeprazole 20mg daily for 6 weeks
  Other Names: DIC; Diclofenac DR; Voltarin
  Arms: Diclofenac
Drug: Meloxicam — meloxicam 7.5mg tablets every 12 hours for 6 weeks; omeprazole 20mg daily for 6 weeks
  Other Names: MLX
  Arms: Meloxicam
Drug: Celecoxib — Celecoxib 200mg capsule every 12 hours for 6 weeks; omeprazole 20mg daily for 6 weeks
  Other Names: CEL
  Arms: Celecoxib

SUMMARY:
This is a 6-week randomized, double-blind trial of 4 different non-steroidal anti-inflammatory drugs in patients with axial spondyloarthritis to compare the change of pain score from baseline at 4 weeks to the change of pain score from baseline at 6 weeks.

DETAILED DESCRIPTION:
Patients with ankylosing spondylitis or axial spondyloarthritis who fulfills the inclusion and exclusion criteria will be randomized into one of the four arms after an initial one week washout period, including: 1) indomethacin 75mg every 12 hours (Q12H); 2) diclofenac 75mg Q12H; 3) meloxicam 7.5mg Q12H; 4) celecoxib 200mg Q12H. The treatment length will be 6 weeks. Primary outcome is the change of pain score from baseline to week 4 and to week 6.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of ankylosing spondylitis (AS) by treating rheumatologists, or a diagnosis of axial spondyloarthritis (axSpA) with a pelvis MRI with significant bone marrow edema on STIR sequences;
* Minimum of 18 years old;
* Are taking NSAIDs on a regular basis for AS or axSpA (defined as more than 20 days in the past month) and willing to withhold medication for one week; or having active symptoms that require initiation of NSAIDs;
* Concomitant anti-rheumatic drugs are allowed, if the dose has been stable for the past three months;
* Have active disease after initial washout period, defined by BASDAI >=4/10, or back pain numerical rating scale (NRS)>=4/10

Exclusion Criteria:

* Patients who have concurrent rheumatic diseases other than AS or axSpA;
* Patients who have oral corticosteroid in the past two weeks; patients who have acute peripheral arthritis;
* Patients with a fibromyalgia score >= 13;
* Patient with extensive cardiac history, history of gastrointestinal bleeding that required blood transfusion, chronic kidney diseases, abnormal liver function tests; or female patients who are pregnant.

Use of low-dose of aspirin (<100mg daily) is allowed in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Runsheng Wang, MD, MHS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a self-controlled study, the objective of the study is to compare the change at week 4 vs. week 6. The participants were randomized into 4 groups getting different drugs, but this is considered as one variable. The study does not intend to compare drug efficacy between arms.
Groups:
- NSAIDs: Diclofenac Delayed Release Oral Tablet 75mg by mouth, every 12 hours for 6 weeks; OR Indomethacin Extended Release Oral Tablet 75mg by mouth, every 12 hours for 6 weeks; OR Meloxicam tablet 7.5mg by mouth, every 12 hours for 6 weeks; OR Celecoxib 200mg capsule by mouth, every 12 hours for 6 weeks
Period: Overall Study
Arm/Group | NSAIDs
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This is a self-controlled study, the objective of the study is to compare the change at week 4 vs. week 6. The participants were randomized into 4 groups getting different drugs, but this is considered as one variable. The study does not intend to compare drug efficacy between arms.
Arm/Group | NSAIDs
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Pain [Median (Full Range); unit: units on a scale] — Pain score by numerical rating score from baseline [scale range: 0 (better) -10 (worse)]
  units on a scale | 6 [3 to 8]
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) [Median (Full Range); unit: units on a scale] — BASDAI by numerical rating score from baseline [scale range: 0 (better) -10 (worse)]
  units on a scale | 4.9 [1 to 7.65]
Bath Ankylosing Spondylitis Function Index (BASFI) [Median (Full Range); unit: units on a scale] — BASFI by numerical rating score from baseline [scale range: 0 (better) -10 (worse)]
  units on a scale | 3.7 [0.4 to 8.4]
ASAS Endorsed Disease Activity Score (ASDAS) [Median (Full Range); unit: units on a scale] | 3.34 [2.03 to 4.79]

OUTCOME MEASURES:

1. Primary Outcome: Change of Pain Score
Description: Change of pain score by numerical rating score from baseline [scale range: 0 (better) -10 (worse)]
Time Frame: Baseline, Week 4, and Week 6
Population: as for baseline characteristics
Measure: Median (Full Range); unit: units on a scale
Groups:
- NSAIDs x 4 Weeks: NSAIDs x 4 weeks
- NSAIDs x 6 Weeks: NSAIDs x 6 weeks
Arm/Group | NSAIDs x 4 Weeks | NSAIDs x 6 Weeks
Number analyzed (Participants) | 9 | 9
units on a scale | -2 [-6 to 2] | -2 [-5 to 0]

2. Secondary Outcome: Change of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: Change of BASDAI by numerical rating score from baseline [scale range: 0 (better) -10 (worse)]
Time Frame: Baseline, Week 4, and Week 6
Population: as for baseline characteristics
Measure: Median (Full Range); unit: units on a scale
Arm/Group | NSAIDs x 4 Weeks | NSAIDs x 6 Weeks
Number analyzed (Participants) | 9 | 9
units on a scale | -1.7 [-6.08 to 0.48] | -2.09 [-5.05 to 0.48]

3. Secondary Outcome: Change of Bath Ankylosing Spondylitis Function Index (BASFI)
Description: Change of BASFI by numerical rating score from baseline [scale range: 0 (better) -10 (worse)]
Time Frame: Baseline, Week 4, and Week 6
Population: as for baseline characteristics
Measure: Median (Full Range); unit: units on a scale
Arm/Group | NSAIDs x 4 Weeks | NSAIDs x 6 Weeks
Number analyzed (Participants) | 9 | 9
units on a scale | -0.8 [-5.8 to 1.7] | -1.2 [-4.2 to 0.4]

4. Secondary Outcome: Change of ASAS Endorsed Disease Activity Score (ASDAS)
Description: Change of ASDAS by numerical rating score from baseline [scale range: 0 (better) -10 (worse)]
Time Frame: Baseline, Week 4, and Week 6
Population: as for baseline characteristics
Measure: Median (Full Range); unit: units on a scale
Arm/Group | NSAIDs x 4 Weeks | NSAIDs x 6 Weeks
Number analyzed (Participants) | 9 | 9
units on a scale | -0.37 [-1.44 to 0.29] | -0.84 [-1.58 to -0.01]

5. Secondary Outcome: Patient Global Assessment of Response to Therapy (PGART)
Description: Likert Scale on whether effective or not.
Time Frame: Week 6
Population: The participants were randomized into 4 groups getting different drugs, but this is considered as one variable. The study does not intend to compare drug efficacy between arms.
Measure: Count of Participants; unit: Participants
Arm/Group | NSAIDs x 6 Weeks
Number analyzed (Participants) | 9
Participants
  Strongly Disagree | 0
  Somewhat Disagree | 0
  Neutral | 2
  Somewhat Agree | 3
  Strongly Agree | 4

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: The participants were randomized into 4 groups getting different drugs, but this is considered as one variable. The study does not intend to compare drug efficacy between arms.
Arm/Group | Celecoxib | Meloxicam | Indomethacin | Diclofenac
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/3 | 1/2 | 2/2 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Celecoxib (N=3) | Meloxicam (N=2) | Indomethacin (N=2) | Diclofenac (N=2)
diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/65/NCT03473665/Prot_SAP_002.pdf